CLINICAL TRIAL: NCT03682471
Title: Long-term, Follow-up Study of Subjects Who Completed Phase III Trials ATX-101-10-16 or ATX-101-10-17 (Sodium Deoxycholate Injection) for the Reduction of Localized Subcutaneous Fat in the Submental Area
Brief Title: Long-term 24-month Follow-up Study on Safety and Maintenance of Efficacy of ATX-101 (Sodium Deoxycholate Injection)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 1403740; 16045 (Other: Company internal); 2011-005026-21 (EudraCT Number); NCT02052622 (obsolete NCT alias)
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Subcutaneous Fat
Keywords: submental fat reduction
MeSH Terms: interventions — Deoxycholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Deoxycholic Acid Injection, 5 mg/mL: Non-treatment observational follow-up study: Participants were previously treated with deoxycholic acid injection, 5 mg/mL in studies ATX-101-10-16 or ATX-101-10-17.
  Interventions: Drug: Deoxycholic acid Injection
- Deoxycholic Acid Injection, 10 mg/mL: Non-treatment observational follow-up study: Participants were previously treated with deoxycholic acid injection, 10 mg/mL in studies ATX-101-10-16 or ATX-101-10-17.
  Interventions: Drug: Deoxycholic acid Injection
- Placebo: Non-treatment observational follow-up study: Participants were previously treated with placebo in studies ATX-101-10-16 or ATX-101-10-17.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deoxycholic acid Injection — Solution for subcutaneous injection.
  Other Names: Kybella
  Groups: Deoxycholic Acid Injection, 10 mg/mL; Deoxycholic Acid Injection, 5 mg/mL
Drug: Placebo — Placebo, 10 mM sodium phosphate, 0.9% [w/v] sodium chloride in water for subcutaneous injection.
  Groups: Placebo

SUMMARY:
The objective of this non-treatment, placebo-controlled, observational, 24-month follow-up study was to evaluate the long-term efficacy and safety of subcutaneous (SC) injections of deoxycholic acid (ATX-101) in the submental area. No treatment was administered in this study. Participants who previously received deoxycholic acid injections in studies ATX-101-10-16 [NCT01305577] or ATX-101-10-17 [NCT01294644] were enrolled in this non-treatment observational follow-up study to further evaluate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any study-related activities are carried out
* Any participant who successfully completed the final visit (visit 7) of a phase 3 clinical trial, ATX-101-10-16 or ATX-101-10-17 for the reduction of submental fat, i.e. subjects must have at least one study treatment administered and have completed the predecessor study up to visit 7
* Willingness to comply with the schedule and procedures of the study

Exclusion Criteria:

* Participants who, since the completion of the prior phase 3 study ATX-101-10-16 or ATX-101-10-17, have had or who are undergoing treatment that may affect the evaluation of the submental area (e.g. - but not limited to - long-term treatment with systemic corticosteroids, liposuction, surgery or other lipolytic treatment in the submental area, treatment with radio frequency, laser procedures, chemical peels, dermal fillers in the neck or chin area or botulinum toxin injections in the neck or chin area)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A subset of participants at selected centers who had successfully completed Phase 3 clinical studies ATX-101-10-16 or ATX-101-10-17 for the reduction of submental fat were enrolled.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2012-02-14 (Actual); Primary Completion 2013-12-13 (Actual); Study Completion 2013-12-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Maintaining Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) 1-Grade Response During the 24 Months of Follow up, i.e. % of Participants who were CR-SMFRS 1-Grade Responders at both LTFU Baseline and at 24-Month Visit | LTFU Baseline (Month 0) to Month 24
  The CR-SMFRS was based on the investigator's clinical evaluation of the participant's chin and neck area using a 5-point ordinal scale (0 to 4) with 0=Absent Submental Convexity: no localized submental fat evident; 1=Mild Submental Convexity: minimal, localized submental fat; 2=Moderate Submental Convexity: prominent, localized submental fat; 3=Severe Submental Convexity; a marked amount of chin fat; and 4=Extreme Submental Convexity: marked, localized submental fat. 1-grade response=At least a 1-grade reduction from original study baseline in the CR-SMFRS assessment.
Percentage of Participants with Maintenance of Response as Assessed by the Subject Satisfaction Rating Scale (SSRS) During the 24 Months of Follow up, i.e. % of Participants who were SSRS Responders at both LTFU Baseline and at 24-Month Visit | LTFU Baseline (Month 0) to Month 24
  For the SSRS, the participant was asked to answer the question: "Considering your appearance in association with your face and chin, how satisfied do you feel with your appearance at the present time?" using a 7-point scale: 0=Extremely dissatisfied, 1=Dissatisfied, 2=Slightly dissatisfied, 3=neither satisfied nor dissatisfied, 4=Slightly satisfied, 5=Satisfied, and 6=Extremely satisfied. SSRS responder was a participant whose response was ≥ 4.

SECONDARY OUTCOMES:
Percentage of Participants Maintaining Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) 2-Grade Response During the 24 Months of Follow up, i.e. % of Participants who were CR-SMFRS 2-Grade Responders at both LTFU Baseline and at 24-Month Visit | LTFU Baseline (Month 0) to Month 24
  The CR-SMFRS was based on the investigator's clinical evaluation of the participant's chin and neck area using a 5-point ordinal scale (0 to 4) with 0=Absent Submental Convexity: no localized submental fat evident; 1=Mild Submental Convexity: minimal, localized submental fat; 2=Moderate Submental Convexity: prominent, localized submental fat; 3=Severe Submental Convexity; a marked amount of chin fat; and 4=Extreme Submental Convexity: marked, localized submental fat. 2- grade response=At least a 2-grade reduction from original study baseline in the CR-SMFRS assessment.
Patient-Reported Submental Fat Impact Scale (PR-SMFIS) | LTFU Baseline (Month 0) to Month 24
  The PR-SMFIS assessed the impact of submental fat on self-perception of 6 emotional and visual characteristics related to the appearance of submental fullness (unhappy, bothered, self-conscious, embarrassed, look older, and look overweight) as evaluated by the participant. Each item was rated on an 11-point numeric scale from 0 to 10. Scores for the 6 items were averaged to generate a PR-SMFIS total scale score ranging from 0 to 10 where low scores reflect a positive impact and high scores reflect a negative impact.
Percentage of Participants Maintaining Composite SMFRS 1-Grade Response During the 24 Months of Follow up, i.e. % of Participants who were Composite SMFRS 1-Grade Responders at both LTFU Baseline and at 24-Month Visit | LTFU Baseline (Month 0) to Month 24
  Participants who had at least a 1-grade reduction in both the CR-SMFRS and PR-SMFRS from the original baseline value in the predecessor study were defined as composite SMFRS-1 responders.
Percentage of Participants with at Least One Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  An adverse event was any undesirable medical occurrence or worsening of an existing condition, irrespective of whether the event was considered treatment-related. A treatment-emergent adverse event was defined as an adverse event with an onset that occurs after receiving treatment.
Percentage of Participants with Treatment-emergent Adverse Events Associated with the Treatment Area (Drug-related) | Up to approximately 24 months
  An adverse event was any undesirable medical occurrence or worsening of an existing condition, irrespective of whether the event was considered treatment-related. A treatment-emergent adverse event was defined as an adverse event with an onset that occurs after receiving treatment.
Percentage of Participants with Treatment-emergent Adverse Events of Special Interest (AESIs) | Up to approximately 24 months
  An adverse event was any undesirable medical occurrence or worsening of an existing condition, irrespective of whether the event was considered treatment-related. A treatment-emergent adverse event was defined as an adverse event with an onset that occurs after receiving treatment. AESIs for this study are common treatment reactions (consistently reported for overall AEs, treatment area-related AEs, or study-drug-related AEs) that were observed in earlier deoxycholic acid injection studies and identified as likely to be related to the injection procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Beta Bowen, Study Director — Allergan
Locations (18):
- Germany (18):
  - Licca Clinical Research Institute, Augsburg
  - Campus Charité Mitte, Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Ruhruniversität Bochum - St. Josef Hospital, Bochum
  - Klinikum Darmstadt, Darmstadt
  - Krankenhaus Dresden- Friedrichstadt Klinik für Dermatologie und Allergologie, Dresden
  - Dr. Beatrice Gerlach, Dresden
  - Klinikum der Johann-Wolfgang Goethe-Universität - Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - Hautarztpraxis Cutanis, Freiburg im Breisgau
  - Praxis Dr. Walker and Dr. Biwer, Ludwigshafen
  - Universitätsklinik Schleswig Holstein, Campus Luebeck, Klinik f. Dermatologie, Lübeck
  - Gemeinschaftsprax is für Dermatologie, Mahlow
  - Ludwig- Maximilians- Universität München, Klinik für Dermatologie und Allergologie, München
  - Germania Campus PraxisKlinik, Münster
  - Praxis Dr. Graefe, Northeim
  - Haut- und Laserzentrum Potsdam, Potsdam
  - Klinik für Dermatologie und Allergologie Klinikum Vest GmbH Recklinghausen, Recklinghausen
  - Hautzentrum am Starnberger See GmbH, Starnberg
  - Dermatologische Privatpraxis, Wuppertal